CLINICAL TRIAL: NCT06720571
Title: Auricular Vagal Neuromodulation Therapy (aVNT) for Enhancing Emotion Regulation, Executive Functions, Hyperphagia, and Quality of Life in Prader-Willi Syndrome: A Multicenter Randomized Controlled Trial
Brief Title: Effects of Transcutaneous Vagus Nerve Stimulation on Emotion Regulation and Executive Functioning in Prader-Willi Syndrome
Acronym: STIM-PRADER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bordeaux (Other)
Collaborators: John Bost Foundation (Unknown); University Hospital, Bordeaux (Other); Hendaye hospital (Unknown); Groupe Hospitalier Pitie-Salpetriere (Other); University Hospital, Toulouse (Other); Prader-Willi Syndrome Association (Other)
Responsible Party: Principal Investigator, Virginie Postal, Researcher and Professor, University of Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A00915-40
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; Vagus nerve stimulation; aVNT; t-VNS; Cognition; Executive functions; Inhibition; Flexibility; Planning; Updating; Emotion regulation; Behavior; Hyperphagia; Quality of life; Depression; Multicenter randomized controlled trial; Caregivers
MeSH Terms: conditions — Prader-Willi Syndrome; Inhibition, Psychological; Emotional Regulation; Behavior; Hyperphagia; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental)
  Interventions: Device: Auricular vagal neuromodulation therapy (aVNT)
- Sham stimulation (Sham Comparator)
  Interventions: Device: Sham Auricular vagal neuromodulation therapy (aVNT)

INTERVENTIONS:
Device: Auricular vagal neuromodulation therapy (aVNT) — The aVNT device used in our study (Parasym ®) consists of a small portable unit connected to stimulation electrodes placed on the left ear. These electrodes deliver painless electrical microcurrents through the skin to stimulate the auricular branch of the vagus nerve (ABVN). The device parameters will be defined in accordance with the recommendations for use of the Parasym ® device and the pilot studies: frequency of 25 Hz, pulse width of 250 µS, and an intensity of 1 mA to 36 mA. Stimulation sessions will last for four hours each day, each of which can be divided into two sessions and conducted over a period of nine months. Patients will adjust the intensity at each session according to their comfort level, starting with a gradual increase until they feel a slight tingling sensation, followed by a decrease until discomfort disappears completely. Stimulation should take place during a relaxing activity but not should not take place during sleep, meals or major physical activity.
  Arms: Active stimulation
Device: Sham Auricular vagal neuromodulation therapy (aVNT) — The sham stimulation control condition will be performed using the same aVNT Parasym® device under similar conditions (four hours a day, seven days a week, for nine months) but with a different location (without afferent vagus nerve fibers) or a control condition integrated into the device.
  Arms: Sham stimulation

SUMMARY:
The STIM-PRADER study aims to assess the effectiveness of auricular vagal neuromodulation therapy (aVNT) on emotional, behavioral, and cognitive domains impaired in Prader-Willi Syndrome (PWS). Currently, no treatment exists that addresses the multiple alterations associated with this rare neurodevelopmental disorder that significantly impact patients and their families. We will investigate the effects of daily, four-hour aVNT stimulation over a nine-month period on (a) emotion regulation, including assessing the persistence of effects following stimulation; (b) executive functions, including inhibition, flexibility, planning, and updating information in memory; (c) hyperphagia; (d) depression; (e) quality of life; (e) and the threshold at which effects on these dimensions can be observed.

We will conduct a longitudinal multicenter parallel randomized controlled single-blind exploratory trial. Twenty-four adults with PWS and 24 caregivers will be randomly assigned to receive either active or sham stimulation under identical conditions (four hours per day, seven days per week over nine months). The primary outcome, focusing on emotional control, will be assessed every two weeks for both participants and caregivers. Secondary outcomes (executive functions, hyperphagia, depression, and quality of life) will be measured at four time points: pre-intervention, at three months, six months, and at nine months.

As this is the first multicenter randomized controlled trial investigating the effects of aVNT as a treatment in PWS patients, we anticipate witnessing improved emotional regulation and reduced eating disorders, along with enhancements in executive functions and quality of life in the active stimulation group. The findings from this project could support the development of broader therapeutic approaches for other conditions in which behavioral disorders and emotional processing deficits affect patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Participant with PWS: Age : ≥ 18 years old; Diagnosis of Prader-Willi syndrome with identified genotype; Intellectual Quotient ≥ 55 measured by WAIS-IV (abbreviated version); Pathological or threshold score on at least one of the BRIEF-A subscales; Adults volunteering and able to comply with study procedures; Signature of informed consent form; Beneficiary of a social security regime
* Caregivers: Caregivers involved in the participant's family, medical or institutional environment; Caregiver who has signed the informed consent form.

Exclusion Criteria:

* Participant with PWS: Untreated and unstabilized psychiatric and/or behavioral disorders (psychological decompensation within the last year); Severe visual or hearing impairment; Untreated sleep apnea syndrome; Epileptic seizures; Previous significative ECG abnormality; Adults with pacemakers or defibrillators; Metal or electronic devices implanted in the head; Participation in other research involving an exclusion period still in progress at inclusion; Score ≥ 30 indicating severe depression (BDI-II self-report questionnaire); Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of emotional control and regulation | Every 2 weeks for 11 months (including 3 times before and post-stimulation)
  The primary outcome measure will focus on assessing emotional control (EC) through a subscale of the BRIEF-A (Behavior Inventory Related to Executive Functions - Adult version).

SECONDARY OUTCOMES:
Evaluation of Behavioral manifestations of executive functioning | 4 times (at 0, 3, 6 and 9 months)
  BRIEF-A (Behavior Inventory Related to Executive Functions - Adult version)
Evaluation of Executive functions | 4 times (at 0, 3, 6 and 9 months)
  Behavioral inhibition will be assessed using a computerized Go/NoGo task and cognitive flexibility with a computerized voluntary alternation task. Planning abilities will be assessed using the BADS Zoo Test (Behavioral Assessment of Dysexecutive Syndrome - BADS). Finally, the ability to update information will be assessed using an adapted computerized N-2-Back task.
Evaluation of Hyperphagia | 4 times (at 0, 3, 6 and 9 months)
  Hyperphagia will be assessed using a scale derived from the Dykens Hyperphagia Questionnaire: the HQ-CT (Hyperphagia Questionnaire for Use in Prader-Willi Syndrome Clinical Trials)
Evaluation of Depression | 4 times (at 0, 3, 6 and 9 months)
  Depression will be assessed using the Depression Self-Report Questionnaire (Beck Depression Inventory - BDI-II)
Evaluation of Quality of life | 4 times (at 0, 3, 6 and 9 months)
  We will assess the quality of life of participants with PWS using the WHOQOL-BREF questionnaire (World Health Organization Quality of Life-BREF)

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Postal, PhD, Principal Investigator — University of Bordeaux
Locations (4):
- France (4):
  - Reference Center of Prader-Willi Syndrome (PRADORT), Bordeaux
  - Reference Center of Prader-Willi Syndrome (CRMR PRADORT), Hendaye
  - Reference Center of Prader-Willi Syndrome (PRADORT), Paris
  - Reference Center of Prader-Willi Syndrome (PRADORT), Toulouse

IPD SHARING:
Plan to Share IPD: Undecided